CLINICAL TRIAL: NCT03833349
Title: The Impact of Three Distinct Exercise Types on Fatigue, Anxiety, and Depression in Parkinson's Disease
Acronym: PDExercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Premier Health (Other)
Collaborators: Parkinson's Disease Foundation (Other); Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 06538
Record Dates: First submitted 2019-02-05; First posted 2019-02-07 (Actual); Last update posted 2020-03-04 (Actual); Status verified 2020-03

CONDITIONS: Parkinson Disease
Keywords: Parkinson's disease; fatigue; anxiety; depression; exercise
MeSH Terms: conditions — Parkinson Disease; Fatigue; Anxiety Disorders; Depression; Motor Activity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Spinning Class (Experimental): Subjects randomly selected for the spinning group will participate in spinning classes, twice a week for six weeks. Subjects will complete questionnaires at screening, each week during the class sessions, and for 1 month follow-up.
  Interventions: Behavioral: Spinning Class
- Yoga Class (Experimental): Subjects randomly selected for the yoga group will participate in yoga classes, twice a week for six weeks. Subjects will complete questionnaires at screening, each week during the class sessions, and for 1 month follow-up.
  Interventions: Behavioral: Yoga Class
- Dance Class (Experimental): Subjects randomly selected for the dance group will participate in dance classes, twice a week for six weeks. Subjects will complete questionnaires at screening, each week during the class sessions, and for 1 month follow-up.
  Interventions: Behavioral: Dance Class

INTERVENTIONS:
Behavioral: Spinning Class — Spinning Class twice a week for six weeks.
  Arms: Spinning Class
Behavioral: Yoga Class — Yoga Class twice a week for six weeks.
  Arms: Yoga Class
Behavioral: Dance Class — Dance Class twice a week for six weeks.
  Arms: Dance Class

SUMMARY:
The purpose of the study is to learn about the impact of exercise on fatigue, anxiety, and depression in Parkinson's disease. It is well established that exercise improves the motor symptoms of Parkinson's disease. However, it is not clear which types of exercise are most beneficial for specific non-motor symptoms.

DETAILED DESCRIPTION:
This is a multi-site trial (12 patients in each site). The investigators are recruiting 24 patients who will be randomized into either a spinning class, yoga class, dance class, or no exercise intervention. Classes will be conducted twice a week for 6 weeks total at times convenient for the patients. Patients will also be asked to complete questionnaires after exercise classes to see if the exercise intervention improves measures of fatigue, anxiety, and depression - and what exercise intervention may be superior. All participants will be asked to complete questionnaires each week and will be asked to wear a "Microsoft exercise band" during the course of the study. Use of the exercise band is optional.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects diagnosed with Idiopathic Parkinson's Disease
2. Age between 18 - 75 years
3. Hoehn and Yahr stage less than or equal to 3
4. Mini-Mental State Exam (MMSE) score of over 23 at screening
5. If subjects are taking any medications for depression, fatigue, or anxiety, regimen must be stable for 8 weeks prior to baseline visit
6. Subjects willing and able to give informed consent

Exclusion Criteria:

1. Subjects with a diagnosis of an atypical Parkinsonism
2. Subjects unwilling or unable to obtain Health Waiver from Primary Care Provider
3. Score of 60 or more on UPDRS III at screening
4. Scores in the 'normal' range on all three study assessments: Beck Depression Index II, Fatigue Severity Scale, and Zung self-rating Anxiety Scale
5. Participation in any of the 3 physical activities more than 3 times in the past for 8 weeks prior to baseline
6. Any other reason that, in the investigator's opinion, would exclude the subject from participation in the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2019-02-11 (Actual); Primary Completion 2019-10-02 (Actual); Study Completion 2019-10-02 (Actual)

PRIMARY OUTCOMES:
Change from baseline, if any, in subjects' Fatigue Severity Scale | screening through study completion, up to 18 weeks
  Subjects will complete the Fatigue Severity Scale at screening and once per week during the exercise class session. Subjects also will receive a follow-up questionnaire to be completed 1 month after the class sessions end. Each item is scored from 1(strongly disagree) to 7(strongly agree).
Change from baseline, if any, in subjects' Zung self-report Anxiety Scale | screening through study completion, up to 18 weeks
  Subjects will complete the Zung self-report Anxiety Scale at screening and once per week during the exercise class session. Subjects also will receive a follow-up questionnaire to be completed 1 month after the class sessions end. Each item is scored from 1(a little of the time) to 4(most of the time).
Change from baseline, if any, in subjects' Beck Depression Inventory II scale | screening through study completion, up to 18 weeks
  Subjects will complete the Beck Depression Inventory II at screening and once per week during the exercise class session. Subjects also will receive a follow-up questionnaire to be completed 1 month after the class sessions end. Each item is scored from 0(Normal) to 3(Severe).

CONTACTS AND LOCATIONS:
Overall Officials: Mary Feldman, DO, Principal Investigator — Premier Health
Locations (2):
- United States (2):
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Premier Health, Dayton, Ohio

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2024 Apr 8;4(4):CD013856. doi: 10.1002/14651858.CD013856.pub3. PMID 38588457
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2023 Jan 5;1(1):CD013856. doi: 10.1002/14651858.CD013856.pub2. PMID 36602886